CLINICAL TRIAL: NCT03420586
Title: Effects of Nitrous Oxide Added at the End of Sevoflurane Anesthesia on Recovery and Postoperative Nausea and Vomiting - a Randomized Clinical Trial (SEVONATE)
Brief Title: Nitrous Oxide Added at the End of Sevoflurane Anesthesia and Recovery
Acronym: SEVONATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital Zadar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01-5623-7/17
Record Dates: First submitted 2018-01-19; First posted 2018-02-05 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2020-08

CONDITIONS: Elective Surgical Procedures; Laparoscopy; Laparotomy; Anesthesia, General; Anesthesia Recovery Period
Keywords: Anesthetics, Inhalation; Anesthesia Recovery Period; Postoperative Nausea and Vomiting; Pain, Postoperative
MeSH Terms: conditions — Respiratory Aspiration; Postoperative Nausea and Vomiting; Pain, Postoperative | interventions — Nitrous Oxide

STUDY DESIGN:
Intervention Model Description: Intervention Model: Parallel Assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects will be randomized into two groups by computer-generated random numbers. Each allocation number will be concealed in an opaque envelope before the start of the surgery and will be revealed 30 min before the end of the operation. Early recovery (eye opening, following verbal commands, time to extubation, orientation to time and place) will be recorded by an anesthesiologist blinded to the anesthesia technique. The same anesthesiologist blinded to the anesthesia technique will collect all postoperative data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nitrous oxide Group (Active Comparator): The nitrous oxide group (GN2O) will receive air in 30% O2 during general anesthesia until the last 30 min of surgery, when 70% N2O in 30% O2 will be administered.
  Interventions: Drug: Nitrous Oxide
- Oxygen Group (No Intervention): The Oxygen group will receive gas carrier mixture consisting of air in 30% O2 during general anesthesia.

INTERVENTIONS:
Drug: Nitrous Oxide — The nitrous oxide group (GN2O) will receive 70% N2O in 30% O2 at the end of surgery.
  Arms: Nitrous oxide Group

SUMMARY:
Addition of nitrous oxide N2O towards the end of prolonged isoflurane anesthesia hastens patients recovery. The hypothesis is that the addition of N2O at the end of prolonged sevoflurane anaesthesia also hastens early recovery without increasing the frequencies and intensity of PONV and improves quality of recovery.

DETAILED DESCRIPTION:
The investigators will include 100 adult patients, American Society of Anesthesiologists (ASA) physical status I-III, who will be scheduled for elective laparotomies or laparoscopic surgeries under sevoflurane anesthesia lasting 120 minutes or longer. After written informed consent participants will be randomized into two groups: GO2 - air in 30% oxygen and GN2O - the same mixture until the last 30 minutes of surgery when 70% N2O in 30% oxygen will be used. General anesthesia will be performed with propofol and fentanyl for anesthesia induction, rocuronium for muscle relaxation and volatile anesthetic sevoflurane for maintenance. The participants will be extubated in the operation room (OR) after they open their eyes and follow commands. Postanesthetic recovery score by Aldrete, Ramsay sedation scale (RSS), and Simplified postoperative nausea and vomiting impact scale score by Myles (PONV ISS) will be used to assess recovery in PACU and surgical ward. Modified Aldrete score assigns a score of 0, 1, or 2 to activity, respiration, circulation, consciousness, and color, giving a maximal score of 10 ( score of 9 indicates recovery sufficient for the patient to be transferred from the PACU). RSS [score 1-6] consists of six levels of sedation [Awake levels: 1, anxious and agitated or restless or both; 2, co-operative, orientated, and tranquil; 3,responds to commands only. Asleep levels are dependent on the response to a light glabellar tap or loud auditory stimulus: 4, a brisk response; 5, a sluggish response; 6, no response]. PONV ISS is the sum of the numerical responses to questions Q1 and Q2 ( Q1: The vomiting or dry-retching count? 0 - 2 or 3 (three or more times); Q2: Severity of nausea - interference with activities of daily living: score 0-3 [0 - not at all, 1-sometimes, 2- often or most of the time, 3 - all of the time] and score ≥5 defines clinically important PONV. Quality of Recovery questionnaire (QoR-40) on the first, second and third postoperative days will be used for assessment of postoperative quality of recovery.The QoR-40 consists of five clinically relevant dimensions: (i) physical comfort (12 items), (ii) emotional state (9 items), (iii) physical independence (5 items), (iv) psychological support (7 items), and (v) pain (7 items). Each item is rated on a five-point Likert scale. The QoR-40 score ranges from 40 (extremely poor quality of recovery) to 200 (excellent quality of recovery). A 100 mm visual analogue scale (VAS) [0= no pain, 10= maximal pain] and the use of postoperative analgesics (opioids/non-opioids: yes or no, quantity in milligrams) shall be used for pain assessment during the first 24 postoperative hours.The sample size for early recovery time (primary endpoint) is based on the results of our recent study. The sample size was calculated on the assumption that 15 (SD 7) min would be needed for early recovery for the GO2 patients and that the GN2O patients would require four minutes less time (11 [SD 5] min). We would need 38 participants in each group for the primary outcome to have a power of 0.8 and an alpha level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, American Society of Anesthesiologists Physical status ASA PS I-III, scheduled for laparotomic and laparoscopic surgery expected to last 2 hours or more who can understand and signed informed consent.

Exclusion Criteria:

* Patients who will be discharged within 72 hours after surgery
* Patients on intensive care within few months before the study enrollment
* Diseases that impair gastric motility (diabetes mellitus, chronic cholecystitis, gastric and intestinal disease, neuromuscular disorders, neuropathies, liver dysfunction)
* Vestibular disease; history of migraine headaches, central nervous system injury
* Renal impairment
* Patients on antihistamines, antipsychotics, contraceptives, steroids within 72 hours before surgery
* Known hypersensitivity to drugs used in the study protocol
* Alcoholism, and/or opioid addiction
* Conditions that can influence the incidence of PONV, postoperative pain or morbidity (e.g., significant intraoperative surgery complications), intraoperative drug allergy, severe intraoperative hypotension, perioperative hypoxia, excessive blood loss, difficult intubation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2021-07-10 (Actual); Study Completion 2021-07-25 (Actual)

PRIMARY OUTCOMES:
Early recovery (awakening) in the operation room (OR) | 15 minutes
  eye opening (in minutes), following verbal commands (in minutes), time to extubation (in minutes ), orientation to time and place (in minutes)

SECONDARY OUTCOMES:
Postoperative nausea and vomiting | 24 hours
  Simplified postoperative nausea and vomiting impact scale:the sum of the numerical responses to questions Q1 and Q2 ( Q1: The vomiting or dry-retching count? 0 -2 or 3 (three or more times); Q2: Severity of nausea - interference with activities of daily living: score 0-3 [0 - not at all, 1-sometimes, 2- often or most of the time, 3- all of the time] ) and score ≥5 defines clinically important PONV.
Quality of recovery | 72 hours
  Quality of Recovery 40 questionnaire on the first, second and third postoperative days: The QoR-40 consists of five clinically relevant dimensions: (i) physical comfort (12 items), (ii) emotional state (9 items), (iii) physical independence (5 items), (iv) psychological support (7 items), and (v) pain (7 items). Each item is rated on a five-point Likert scale. The QoR-40 score ranges from 40 (extremely poor quality of recovery) to 200 (excellent quality of recovery).
Postoperative pain | 24 hours
  Visual analogue scale VAS pain score [a 100 mm visual analogue scale (VAS) 0= no pain, 10= maximal pain]

OTHER OUTCOMES:
Postoperative sedation | 2 hours
  Ramsay Sedation Scale [score 1-6] consists of six levels of sedation [Awake levels: 1, patient anxious and agitated or restless or both; 2, patient co-operative, orientated, and tranquil; 3, patient responds to commands only. Asleep levels are dependent on the patient's response to a light glabellar tap or loud auditory stimulus: 4, a brisk response; 5, a sluggish response; and 6, no response].
Postoperative nausea and vomiting | 24 hours
  The use of rescue antiemetics (yes/no and quantity in milligrams)
Postoperative pain | 24 hours
  The use of analgesics (opioids/nonopioids:yes/no and quantity in milligrams)
Readiness for Discharge from the Postanesthesia Care Unit (PACU) | 2 hours
  Modified Aldrete score: Activity - able to move voluntarily or on command: 2 - four extremities ; 1- two extremities ; 0- extremities 0; Respiration: 2 - able to deep breathe and cough freely , 1 - dyspnea, shallow or limited breathing , 0 - apneic. Circulation - blood pressure , BP of preanesthetic level: 2 - BP ± 20 mm; 1 - BP ± 20-50 mm; 0 - BP ± 50 mm. Consciousness: 2 fully awake;1 arousable on calling; 0 not responding.O2 saturation : 2 - able to maintain O2 saturation >92% on room air; 1- needs O2 inhalation to maintain O2 saturation >90%; 0 - O2 saturation <90% even with O2 supplementation. A score 9 and more = Ready for Discharge from the Postanesthesia Care Unit

CONTACTS AND LOCATIONS:
Overall Officials: Tatjana Simurina, MD, PhD, Principal Investigator — GH Zadar, Dpt. of Anesthesiology and Intensive Care Medicine; Boris Mraovic, Prof, MD, Principal Investigator — Anesthesiology & Parioperative Medicine School of Medicine, University of Missouri, Columbia, US
Locations (1):
- General Hospital Zadar, Zadar, Croatia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mraovic B, Simurina T, Gan TJ. Nitrous oxide added at the end of isoflurane anesthesia hastens early recovery without increasing the risk for postoperative nausea and vomiting: a randomized clinical trial. Can J Anaesth. 2018 Feb;65(2):162-169. doi: 10.1007/s12630-017-1013-y. Epub 2017 Nov 17. PMID 29150782
- [Background] Peyton PJ, Wu CY. Nitrous oxide-related postoperative nausea and vomiting depends on duration of exposure. Anesthesiology. 2014 May;120(5):1137-45. doi: 10.1097/ALN.0000000000000122. PMID 24401771
- [Background] Myles PS, Weitkamp B, Jones K, Melick J, Hensen S. Validity and reliability of a postoperative quality of recovery score: the QoR-40. Br J Anaesth. 2000 Jan;84(1):11-5. doi: 10.1093/oxfordjournals.bja.a013366. PMID 10740540
- [Background] Myles PS, Hunt JO, Nightingale CE, Fletcher H, Beh T, Tanil D, Nagy A, Rubinstein A, Ponsford JL. Development and psychometric testing of a quality of recovery score after general anesthesia and surgery in adults. Anesth Analg. 1999 Jan;88(1):83-90. doi: 10.1097/00000539-199901000-00016. PMID 9895071
- [Background] Myles PS, Wengritzky R. Simplified postoperative nausea and vomiting impact scale for audit and post-discharge review. Br J Anaesth. 2012 Mar;108(3):423-9. doi: 10.1093/bja/aer505. Epub 2012 Jan 29. PMID 22290456
- [Background] Agoliati A, Dexter F, Lok J, Masursky D, Sarwar MF, Stuart SB, Bayman EO, Epstein RH. Meta-analysis of average and variability of time to extubation comparing isoflurane with desflurane or isoflurane with sevoflurane. Anesth Analg. 2010 May 1;110(5):1433-9. doi: 10.1213/ANE.0b013e3181d58052. PMID 20418303
- [Background] Jones PM, Bainbridge D, Chu MWA, Fernandes PS, Fox SA, Iglesias I, Kiaii B, Lavi R, Murkin JM. Comparison of isoflurane and sevoflurane in cardiac surgery: a randomized non-inferiority comparative effectiveness trial. Can J Anaesth. 2016 Oct;63(10):1128-1139. doi: 10.1007/s12630-016-0706-y. Epub 2016 Jul 27. PMID 27465213